CLINICAL TRIAL: NCT03343600
Title: A Randomization, Double Blind, Multicenter Phase II Clinical Trial to Evaluate the Imatinib for Prophylaxis of CMV Infection After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Imatinib for Cytomegalovirus Prophylaxis and Treatment After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial is terminated due to the extremely low recruitment rate.
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Far Eastern Memorial Hospital (Other); Tri-Service General Hospital (Other); National Cheng-Kung University Hospital (Other); Hualien Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201707076MIPB
Record Dates: First submitted 2017-09-27; First posted 2017-11-17 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Patients Who Have Received Allo-HSCT
MeSH Terms: interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imatinib (Experimental): Imatinib (100 mg/tablet) 2# per day till D+100 after allo-HSCT or prophylaxis failure.
  Interventions: Drug: Imatinib
- Placebo (Placebo Comparator): Placebo 2# per day till D+100 after allo-HSCT or prophylaxis failure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Imatinib — Imatinib 100 mg/tablet, 2 tablets daily
  Arms: Imatinib
Drug: Placebo — Placebos 2 tablets daily
  Arms: Placebo

SUMMARY:
This study aim at examining whether blocking platelet-derived growth factor receptor-α by imatinib lowers the risk of post-allogeneic hematopoietic stem cell transplantation CMV infection.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multicenter phase II clinical trial. In the trial, post-allo-HSCT patients with signs of bone marrow engraftment and without evidence of CMV reactivation will be enrolled. All enrolled patients will be monitored for their blood CMV DNA copy numbers by Q-PCR and safety throughout the trial. In addition to their routine post-allo-HSCT care, eligible patients will receive imatinib (100mg/tablet, 2 tablets daily) or placebo (2 tablets daily) administration after myeloid engraftment (defined as absolute neutrophil count higher than 500 for three consecutive days). While receiving the trial therapy, patients will have a regular CMV surveillance every week by the quantification of plasma CMV DNA copies. During the administration of the investigational drugs, other concomitant anti-CMV prophylaxis treatments are prohibited. When a patient has any signs suggesting CMV infection that the treating physician determines that an anti-CMV therapy is indicated, the patient will be defined as failure of prophylaxis for the efficacy evaluation. Whether the conventional anti-CMV therapy is started or not, the investigational drugs with imatinib or placebo will be continued till at least Day+100 unless the patient is defined as prophylaxis failure or withdraws from the study including personal reasons, early mortality, disease recurrence after transplantation, pregnancy, or the investigator decides that the subject should be withdrawn for safety reasons or physical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (Age ≧ 20) who received the first allo-HSCT are eligible;
* Patients with underlying disease of acute leukemia in morphological remission, or myelodysplastic syndrome;
* Received allo-HSCT with HLA-matched sibling or unrelated donors (at least 8/8 match for HLA-A/B/C/DR);
* Evidence of post-transplantation neutrophil engraftment: absolute neutrophil count > 500/mm3 for at least 3 consecutive days;
* No detectable CMV infection before study enrollment: negative plasma CMV DNA surveillance within passing 2 weeks;
* No previous post-transplantation anti-CMV therapy and no planned prophylactic anti-CMV therapy;
* The patients has the ability to swallow tablets

Exclusion Criteria:

* They have renal insufficiency: serum creatinine > 2.5 mg/dL;
* They have hepatic dysfunction: serum alanine or aspartate aminotransferase levels of > 5 times the upper limit of the normal range or a serum total bilirubin of > 3 mg/dL;
* Patients with history of HIV infection;
* Unstable post-BMT condition or other medical condition deemed not appropriate to be included to this study as judged by investigator;
* Life expectancy less than 3 months;
* Unwillingness or unable to give consent;
* Patients with diseases that are positive for t(9;22) or BCR-ABL fusion gene.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants free from initiating conventional anti-CMV treatment by Day+100 after allo-HSCT. | From first dosing to 100 days after allo-HSCT (Day+100)
  Investigator determined whether anti-CMV treatment is needed or not based on clinical judgment no matter therapeutic or preemptive treatment. Symptomatic CMV infection or CMV organ disease was defined as described by Ljungman et al., 2002.

SECONDARY OUTCOMES:
Number of treatment-related adverse events (AE) by Day+100 after allo-HSCT. | From first dosing to 100 days after allo-HSCT (Day+100)
  Safety profile will be evaluated according to treatment-related adverse events (AE) per CTCAE 4.03 version.
Time to onset of CMV reactivation defined by peripheral blood CMV copies by Day+100 after allo-HSCT. | From first dosing to 100 days after allo-HSCT (Day+100)
  The peripheral blood CMV DNA copy numbers (copies/mL) were determined using a commercial kit with PCR method following its protocol. The CMV copy numbers are monitored on a weekly basis.
Time to onset of CMV disease diagnosed by investigator by Day+100 after allo-HSCT. | From first dosing to 100 days after allo-HSCT (Day+100)
  The diagnosis of CMV disease is based on clinical practice and the invasive procedure was encouraged to make the definite diagnosis. The reference to CMV organ disease definition was described by Ljungman et al., 2002.
Number of participants who had progressive hematological disease within 6 months after allo-HSCT. | 6 months post-transplant
  Defined as any subject that is known to have a progressive hematological disease.
Number of participants who died within 6 months after allo-HSCT. | 6 months post-transplant
  Defined as any subject that is known to be dead.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Ting Lin, MD, Principal Investigator — National Taiwan University Hospital
Locations (5):
- Taiwan (5):
  - Tzu Chi General Hospital, Hualien City
  - Far Eastern Memorial Hospital, New Taipei City
  - National Cheng Kung Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei